CLINICAL TRIAL: NCT00379522
Title: A Multicenter, Randomized, Controlled Trial Assessing Arginine Vasopressin Versus Saline Placebo in Refractory Traumatic Hemorrhagic Shock Patients (VITRIS-study)
Brief Title: Vasopressin in Traumatic Hemorrhagic Shock Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Volker Wenzel (Other)
Responsible Party: Sponsor-Investigator, Volker Wenzel, Prof. Dr., Medical University Innsbruck
Organization: Medical University Innsbruck (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Vitris
Record Dates: First submitted 2006-09-21; First posted 2006-09-22 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Shock; Hypovolemia; Hemorrhagic Shock
Keywords: hemorrhagic; shock; traumatic; shock treatment; vasopressin; Circulatory Collapse; Hypovolemic Shock
MeSH Terms: conditions — Shock; Hypovolemia; Shock, Hemorrhagic; Diabetes Insipidus | interventions — Vasopressins; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vasopressin (Active Comparator): Vasopressin, 10 I.U./4 ml, Solution for Injection
  Interventions: Drug: Vasopressin
- Saline (Placebo Comparator): Saline placebo 4 ml, Solution for Injection
  Interventions: Drug: Saline placebo

INTERVENTIONS:
Drug: Vasopressin — 10 minutes after standard shock treatment 10 IU arginine vasopressin will be injected; if shock persists for 5 minutes, another 10 IU arginine vasopressin will be injected; after 5 minutes persisting shock, the last 10 IU arginine vasopressin will be injected; Total duration: approx. 15 minutes; Dose per intravenous injection: 10 IU; max. dose: 30 IU arginine vasopressin
  Other Names: Pressyn; CPREssin; Pitressin
  Arms: Vasopressin
Drug: Saline placebo — Placebo for arginine vasopressin
  Other Names: Kochsalz; Saline
  Arms: Saline

SUMMARY:
The purpose of the present trial is therefore to assess effects of arginine vasopressin vs. saline placebo on hospital admission rate (primary end point), as well as hemodynamic variables, fluid resuscitation requirements and hospital discharge rate (secondary study end points) in presumed traumatic hemorrhagic shock patients with a systolic arterial blood pressure <90 mm Hg after 10 min of standard shock treatment. Accordingly, the study reflects an add-on design to standard traumatic shock therapy.

The hypothesis is that both arginine vasopressin and saline placebo have comparable effects on hemodynamic variables, fluid resuscitation requirements, and hospital admission and discharge rate. The alternative hypothesis is that arginine vasopressin has more beneficial effects on hemodynamic variables, fluid resuscitation requirements, and hospital admission and discharge rate than saline placebo.

DETAILED DESCRIPTION:
The study will be designed as a multicenter, randomized, placebo-controlled clinical trial with blinded assessment of the outcome in a study network with helicopter emergency medical service units in Austria, Germany, Switzerland, Italy, Czech Republic and the Netherlands.

The protocol, information and consent procedure will be approved by the institutional review board of each participating center. Since this is a study randomizing unconscious patients who are unable to give informed consent at the time of randomization (§43a Emergency study), the requirement of informed consent is planned to be waived in accordance with the ethical standards of national legislation in Germany, Austria, Switzerland, Italy, Czech Republic and the Netherlands and the guidelines for good clinical practice of the European Agency for the Evaluation of Medicinal products. Depending on the patient's outcome, either the surviving patient, or the patient's family in case of death of the patient or in case that the patient survives but remains mentally handicapped will be informed about the trial (see appendix for patient information sheet); the protocol specifies that if there are any objections, the patient will be withdrawn from the study.

Treatment assignments of blinded study drugs will be randomly generated by computer in blocks of two, with stratification according to center. Before the start of the trial, staff at participating centers will be informed about the rationale of the protocol and the study; participating centers will be subsequently contacted and visited to ensure proper enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adult trauma patients presenting with presumed traumatic hemorrhagic shock (systolic arterial blood pressure <90 mm Hg) that does not respond to the first 10 min of standard shock treatment [endotracheal intubation, crystalloid-, colloid-, and hypertonic saline (up to 4 ml/kg) fluid resuscitation, and catecholamine (ephedrine, phenylephrine, norepinephrine, epinephrine) vasopressors].

Exclusion Criteria:

* Terminal illness
* No intravenous access
* Age < 18 years
* Injury > 60 min before randomization
* Known pregnancy
* Cardiac arrest before randomization
* Presence of a do-not-resuscitate order
* Untreated tension pneumothorax
* Untreated cardiac tamponade
* Participation in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Primary end point will be hospital admission rate | time from trauma to hospital admission

SECONDARY OUTCOMES:
Hemodynamic variables | time from trauma to hospital discharge
Fluid resuscitation requirements | time from trauma to hospital discharge
Hospital discharge rate | time from trauma to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Volker Wenzel, M.Sc., M.D., Study Chair — Innsbruck Medical University, Dep. for Anaesthesia and Crit. Care Management
Locations (14):
- Austria (8):
  - HEMS Ybbsitz / Hospital Amstetten, Amstetten, Lower Austria
  - Hospital Krems, Krems, Lower Austria
  - Hospital Wiener Neustadt, Wiener Neustadt, Lower Austria
  - Hospital Salzburg, Salzburg, Salzburg
  - Medical University of Graz, Graz, Styria
  - Medical University of Innsbruck, Innsbruck, Tyrol
  - Hospital Linz, Linz, Upper Austria
  - HEMS Suben / Landeskrankenhaus Schärding, Schärding, Upper Austria
- Germany (6):
  - University Hospital of Dresden, Dresden
  - University Hospital of Goettingen, Göttingen
  - University Hospital of Mannheim, Mannheim
  - BG-Unfallklinik Murnau, Murnau am Staffelsee
  - Ev. Jung-Stilling-Krankenhaus, Siegen
  - Bundeswehrkrankenhaus Ulm, Ulm

REFERENCES:
- [Background] Krismer AC, Wenzel V, Voelckel WG, Innerhofer P, Stadlbauer KH, Haas T, Pavlic M, Sparr HJ, Lindner KH, Koenigsrainer A. Employing vasopressin as an adjunct vasopressor in uncontrolled traumatic hemorrhagic shock. Three cases and a brief analysis of the literature. Anaesthesist. 2005 Mar;54(3):220-4. doi: 10.1007/s00101-004-0793-y. PMID 15605286
- [Background] Schummer W, Schummer C, Fuchs J. [Vasopressin]. Anaesthesist. 2005 Jul;54(7):707-8. doi: 10.1007/s00101-005-0854-x. No abstract available. German. PMID 15843908
- [Background] Tsuneyoshi I, Onomoto M, Yonetani A, Kanmura Y. Low-dose vasopressin infusion in patients with severe vasodilatory hypotension after prolonged hemorrhage during general anesthesia. J Anesth. 2005;19(2):170-3. doi: 10.1007/s00540-004-0299-4. PMID 15875138
- [Background] Raedler C, Voelckel WG, Wenzel V, Krismer AC, Schmittinger CA, Herff H, Mayr VD, Stadlbauer KH, Lindner KH, Konigsrainer A. Treatment of uncontrolled hemorrhagic shock after liver trauma: fatal effects of fluid resuscitation versus improved outcome after vasopressin. Anesth Analg. 2004 Jun;98(6):1759-1766. doi: 10.1213/01.ANE.0000117150.29361.5A. PMID 15155342
- [Background] Stadlbauer KH, Wenzel V, Krismer AC, Voelckel WG, Lindner KH. Vasopressin during uncontrolled hemorrhagic shock: less bleeding below the diaphragm, more perfusion above. Anesth Analg. 2005 Sep;101(3):830-832. doi: 10.1213/01.ANE.0000175217.55775.1C. No abstract available. PMID 16115999
- [Background] Stadlbauer KH, Wagner-Berger HG, Raedler C, Voelckel WG, Wenzel V, Krismer AC, Klima G, Rheinberger K, Nussbaumer W, Pressmar D, Lindner KH, Konigsrainer A. Vasopressin, but not fluid resuscitation, enhances survival in a liver trauma model with uncontrolled and otherwise lethal hemorrhagic shock in pigs. Anesthesiology. 2003 Mar;98(3):699-704. doi: 10.1097/00000542-200303000-00018. PMID 12606914
- [Background] Voelckel WG, Raedler C, Wenzel V, Lindner KH, Krismer AC, Schmittinger CA, Herff H, Rheinberger K, Konigsrainer A. Arginine vasopressin, but not epinephrine, improves survival in uncontrolled hemorrhagic shock after liver trauma in pigs. Crit Care Med. 2003 Apr;31(4):1160-5. doi: 10.1097/01.CCM.0000060014.75282.69. PMID 12682488
- [Derived] O'Callaghan DJ, Gordon AC. What's new in vasopressin? Intensive Care Med. 2015 Dec;41(12):2177-9. doi: 10.1007/s00134-015-3849-3. Epub 2015 May 7. No abstract available. PMID 25947955
- See also: Study Homepage — http://www.vitris.at